CLINICAL TRIAL: NCT00444509
Title: A Double-blind, Placebo-controlled, Crossover Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single Dose Dry Powder GW685698X Containing Magnesium Stearate in Subjects With Mild to Moderate Asthmatic Patients
Brief Title: Single Dose GW685698X Magnesium Stearate Study In Asthmatic Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: HZA108799
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Asthmatic Patients
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): Subjects will receive GW685698X 800 microgram (mcg) single inhaled dose via a DISKUS inhaler. There will be a wash-out period of at least 5 days between doses.
  Interventions: Drug: GW685698X; Drug: GW685698X containing magnesium stearate
- Treatment 2 (Experimental): Subjects will receive GW685698X 800 mcg containing magnesium stearate inhaled dose via a DISKUS inhaler. There will be a wash-out period of at least 5 days between doses.
  Interventions: Drug: GW685698X; Drug: GW685698X containing magnesium stearate

INTERVENTIONS:
Drug: GW685698X — GW685698X will available with a unit dose strength of 400 mcg that will be inhaled via DISKUS
Drug: GW685698X containing magnesium stearate — GW685698X containing magnesium stearate will available with a unit dose strength of 400 mcg that will be inhaled via DISKUS

SUMMARY:
This is a single centre, randomised, double blind, two-way crossover study, to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of inhaled dry powder GW685698X (800?g) containing magnesium stearate. Magnesium stearate is an excipient added to improve the physical stability of inhaled dry powder formulations. Male and female patients with mild/moderate asthma will be randomised to determine which order they receive a single inhaled administration of GW685698X (800?g) with and without magnesium stearate. There will be a wash-out period of at least 5 days between doses.

ELIGIBILITY:
Inclusion criteria:

* Clinically stable persistent mild/moderate asthma within the 4 weeks preceding the screening visit,
* screening pre-bronchodilator FEV1 >or=60 % predicted,demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of >or= 12.0% over the max of the three screening measures and an absolute change of

  >or= 200 mL within 30 minutes following a single 400 mcg salbutamol dose, male or female (of non child bearing potential or meet the contraception criteria),
* BMI 19-31 kg/m2,
* Non-smoker,
* refrains from use of prohibited medication within the specified timeframes

Exclusion criteria:

* Pregnant or nursing females
* History of life threatening asthma
* Subjects who are unable to stop taking protocol defined prohibited medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02-17 (Actual); Primary Completion 2007-04-09 (Actual); Study Completion 2007-04-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Vital signs: for 48 hours 12-lead ECG including QT, QTc, PR and QRS intervals for 48 hours PEFR, FEV1 for 48 hours Laboratory safety tests (clinical chemistry, haematology, urinalysis) at predose Adverse events for 46 days | Vital signs: for 48 hours

SECONDARY OUTCOMES:
Plasma GW685698X concentrations and pharmacokinetic parameters (AUC, Cmax, t1/2, tmax) following single inhaled doses in mild/moderate asthmatic patients for 48 hours. Weighted mean serum cortisol (0-24 h) on Day 1. | following single inhaled doses in mild/moderate asthmatic patients for 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study HZA108799 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/HZA108799?search=study&search_terms=HZA108799#rs
- Available data/document: Informed Consent Form: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA108799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register